CLINICAL TRIAL: NCT04382040
Title: A Phase II, Controlled Clinical Study Designed to Evaluate the Effect of ArtemiC in Patients Diagnosed With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MGC Pharmaceuticals d.o.o (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MGC-006
Record Dates: First submitted 2020-05-07; First posted 2020-05-11 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; Corona Virus Infection; SARS-CoV 2; Coronavirus; Coronavirus Infection
Keywords: Coronavirus; COVID-19; Intervention Study
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a manner of 2:1 for study drug (ArteminC) and Standard of Care to Placebo and Standard of Care.
  Patient study period will last 2 weeks. During this time, patients will be monitored for adverse events.
  There will be a follow up period (until hospital discharge) in order to check side effects and study drug efficacy
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ArtemiC (Experimental): Active study treatment + Standard care
  Interventions: Drug: ArtemiC
- PLACEBO (Placebo Comparator): Placebo + Standard care
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ArtemiC — Treatment will be sprayed orally twice a day for the first 2 days in the treatment period
  Arms: ArtemiC
Drug: Placebo — Treatment will be sprayed orally twice a day for the first 2 days in the treatment period
  Arms: PLACEBO

SUMMARY:
Agent Name and Study Duration

ArtemiC is a medical spray comprised of Artemisinin (6 mg/ml), Curcumin (20 mg/ml), Frankincense (=Boswellia) (15 mg/ml) and vitamin C (60 mg/ml) in micellar formulation for spray administration.

Patients will receive up to 6 mg Artemisinin, 20 mg Curcumin, 15 mg Frankincense and 60 mg vitamin C given daily as an add-on therapy (in addition to standard care) in two divided doses, on Days 1 and 2.

Patients will be randomized in a manner of 2:1 for study drug (ArteminC) and Standard of Care to Placebo and Standard of Care.

Patient follow-up will last 2 weeks. During this time, patients will be monitored for adverse events.

Additional time will be required for follow up (until hospital discharge) in order to check side effects and study drug efficacy.

Placebo, composed of the same solvent but without active ingredients, will be given in the placebo group as add-on therapy, 2 times a day, on Days 1 and 2.

Overall rationale A preparation of ArtemiC, comprising Artemisinin, Curcumin, Boswellia, and Vitamin C, is proposed as a treatment for the disease associated with the novel corona virus SARS-CoV-2. It is readily available in light of its status as a food supplement. This initiative is presented under the urgent circumstances of the fulminant pandemic caused by this lethal disease, which is known as COVID-19 and has spread across the globe causing death and disrupting the normal function of modern society. The grounds for the proposal are rooted in existing knowledge on the components and pharmacological features of this formulation and their relevance to the current understanding of the disease process being addressed.

Leading among these considerations are well established immuno-modulatory activities of the active ingredients as established in vitro and in vivo and published over the years. These activities as apparent, for example, in diminishing activity of TNF alpha and IL-6 levels are acknowledged to be relevant to the pathophysiology processes involved in the progressive form of COVID-19. The active agents have in addition prominent anti-oxidant, anti-inflammatory as well as anti-aggregant and anti-microbial activities.

Based on these activities and observations in animal models, together with clinical experience of the separate ingredients and in various combinations in other contexts it is proposed to evaluate their effect in the context of COVID-19.

Study Purpose This study is designed to evaluate the safety and efficacy of ArtemiC on patients diagnosed with COVID-19.

Methodology 50 adult patients who suffer from COVID-19 infection studied in parallel groups treated with active agent or placebo as add on to standard care.

Safety will be assessed through collection and analysis of adverse events, blood and urine laboratory assessments and vital signs.

DETAILED DESCRIPTION:
STUDY OBJECTIVES This study is designed to evaluate the safety and efficacy of ArtemiC on patients diagnosed with COVID-19.

STUDY TREATMENT AND DESIGN 50 adult patients who suffer from COVID-19 infection, and do not participant in any other clinical trial.

Patient must agree to not participate in any new clinical study during the study duration.

ArtemiC is a medical spray combined of Artemisinin (6 mg/ml), Curcumin (20 mg/ml), Frankincense (15 mg/ml) and vitamin C (60 mg/ml) in spray administration.

It has a current status as a food supplement. Patients will receive up to 12 mg Artemisinin, 40 mg Curcumin, 30 mg Frankincense and 120 mg vitamin C in 2ml as a total maximum dose, given as add-on therapy, comprised of 2 daily doses of 0.5 ml each, on Days 1 and 2. Each dose contains 0.5 ml (total 1 ml daily dose), which is equal to 5 pushes on the spray bottle.

Placebo, composed of the same solvent but without active ingredients, will be given as add-on therapy in the placebo group, 2 times a day, on Days 1 and 2.

Patients will be randomized in a manner of 2:1 for study drug (ArteminC) and Standard of Care to Placebo and Standard of Care.

The study will last 2 weeks. During this time, patients will be monitored for adverse events.

Additional time will be required for follow up (until hospital discharge) in order to check side effects and study drug efficacy.

STUDY PROCEDURES

Evaluation of the effect of oral administration of the study drug will be assessed by determining the clinical and laboratory tests as summarized below:

Biochemistry Blood Test: Sodium (Na), Potassium (K), Chloride (Cl), Creatinine, Glucose, Urea, Albumin, Calcium total, Alkaline Phosphatase (ALP), ALT, AST, Total Bilirubin, Direct Bilirubin, LDH, Total Protein, Uric Acid, CRP, and Lipid Profile (including Total Cholesterol, HDL, LDL, Triglycerides), D-dimer, ESR as well as Troponin as required.It will be performed per institutional schedule.

Hematology Blood Test: complete CBC. It will be performed per institutional schedule.

Vital signs: blood pressure, pulse, weight, height, temperature. It will be performed per institutional schedule.

Women of childbearing potential must undergo a urine pregnancy test. Physical examination: It will be performed per institutional schedule. All the above measurements will be performed by the hospital staff, not necessarily by the principal investigator or the sub-investigators.

Day 1 Prior to engaging in any study procedures, the subject must meet the inclusion/exclusion criteria by history (which includes a declination), and review and sign an ICF. Following procedures will be performed during the visit -

* Inclusion/Exclusion criteria evaluation
* ICF
* Medical history
* Concomitant medication
* Physical examination
* Vital signs
* Urine pregnancy test (if relevant)
* Test for detection of COVID-19
* Hematology blood test
* Biochemistry blood test
* Randomization (2:1 for study drug (ArteminC) and Standard of Care to Placebo and Standard of Care) and study drug administration

Day 2

* Concomitant medication
* Adverse Events assessment
* Physical examination
* Vital signs
* Hematology blood test
* Biochemistry blood test
* Study drug administration

Days 3-14

* Concomitant medication
* Adverse Events assessment
* Physical examination-is per institutional schedule
* Vital signs- is per institutional schedule
* Hematology blood test- is per institutional schedule
* Biochemistry blood test- is per institutional schedule

Follow up - Hospital Discharge

* Concomitant medication
* Adverse Events assessment
* Physical examination
* Vital signs
* Test for detection COVID-19
* Hematology blood test
* Biochemistry blood test

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed SARS-CoV-2 infection.
2. Hospitalized COVID-19 patient in stable moderate condition (i.e., not requiring ICU admission).
3. Subjects must be under observation or admitted to a controlled facility or hospital (home quarantine is not sufficient).

Exclusion Criteria:

1. Tube feeding or parenteral nutrition.
2. Patients who are symptomatic and require oxygen (Ordinal Scale for Clinical Improvement score >3) at the time of screening.
3. Respiratory decompensation requiring mechanical ventilation.
4. Uncontrolled diabetes type 2.
5. Autoimmune disease.
6. Pregnant or lactating women.
7. Any condition which, in the opinion of the Principal Investigator, would prevent full participation in this trial or would interfere with the evaluation of the trial endpoints.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Time to clinical improvement, defined as a national Early Warning Score 2 (NEWS2) of </= 2 Maintained for 24 Hours in comparison to routine treatment | 24 hours
  patient will be assessed using a scoring table for changes in clinical signs
Percentage of participants with definite or probable drug related adverse events | 14 days
  Adverse events caused by the study drug will be assessed

SECONDARY OUTCOMES:
Time to negative COVID-19 PCR | 14 days
Proportion of participants with normalization of fever and oxygen saturation through day 14 since onset of symptoms | 14 days
COVID-19 related survival | 14 days
Incidence and duration of mechanical ventilation | 14 days
Incidence of Intensive Care Init (ICU) stay | 14 days
Duration of ICU stay | 14 days
Duration of time on supplemental oxygen | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Rubi Zomer, Study Director — MGC Pharmaceuticals
Locations (4):
- Mahatma Gandhi Mission Medical College and Hospital, Aurangabad, Maharashtra, India
- Israel (3):
  - Hillel Yaffe Medical Center, Hadera, Haifa District
  - Nazareth Hospital EMMS, Nazareth, North
  - Rambam Health Care Campus, Haifa

IPD SHARING:
Plan to Share IPD: No